CLINICAL TRIAL: NCT04953091
Title: Evaluation du Test " Sofia SARS Antigen FIA Assay " Dans le Cadre du dépistage de la COVID-19
Brief Title: Evaluation of the Sofia SARS Antigen FIA Assay for COVID-19
Acronym: ESADEC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ESADEC ( 29BRC21.0117)
Record Dates: First submitted 2021-07-06; First posted 2021-07-07 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-04

CONDITIONS: SARS-CoV2 Infection
Keywords: SARS-CoV2 Infection; Assessment; EIA; Diagnosis
MeSH Terms: conditions — COVID-19; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluating the performance of the Sofia SARS Antigen FIA

DETAILED DESCRIPTION:
RT-PCR is the reference technique for the diagnosis of COVID-19, as recommended by WHO, ECDC and the HAS College.

Serological tests to identify antibodies developed by the immune system following infection with SARS-CoV-2 are not currently recommended as a first-line test for the initial diagnosis of COVID-19. However, they can be used in cases of negative RT-PCR and suggestive clinical presentation, or as a salvage test when RT-PCR could not be performed within 7 days of symptom onset.

Antigenic tests for the detection of SARS-CoV-2 can be used as a first-line test on nasopharyngeal swabs up to and including 4 days after the onset of symptoms. From the 5th day, only detection by gene amplification is indicated. Given their excellent specificity and the current pandemic situation, it is not necessary to confirm positives with a gene amplification test.

However, it is recommended to perform a gene amplification test when the antigenic test result is negative or uninterpretable in symptomatic patients older than 65 years or with at least one risk factor for severe COVID-19.

For contact persons detected in isolation or in clusters, it is also possible to use antigenic tests in the following cases

* as soon as possible and then at 7 days for high-risk contacts (within the same household as an infected patient) ;
* 7 days after exposure for other contacts (low risk).

Given the rapidity of antigenic test results (15 to 30 minutes), the good performance of the Sofia SARS Antigen FIA test in target populations and its traceability, it could be used as a first-line test in emergency rooms and screening centers and thus have a positive impact on the management of ambulatory patients and, by corollary, on viral transmission.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (> or = 18 years of age)
* Patient with symptoms of COVID-19 (Rhinitis, throat pain, nasal congestion or other signs of local manifestation of the disease in the upper respiratory tract, including loss of taste, with or without additional systemic symptoms such as fatigue, fever, muscle pain...) whose health condition does not require hospitalization (mild to moderate disease)
* Patient with these symptoms for 5 days or less with a median of 3 to 4 days.
* Patient with consent to participate in the study

Exclusion Criteria:

* Patient with an age below 18 years
* Patient under legal protection (guardianship, curatorship)
* Patient without upper respiratory tract symptoms
* Patients with symptoms for more than 5 days
* Patient with previous COVID-19 diagnosed by RT-PCR
* Patient vaccinated against SARS-CoV-2 (1 or 2 injections)
* Hospitalized patient
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two nasopharyngeal swabs will be taken per included patient. One will be analyzed by RT-PCR in the virology laboratory, the other will be analyzed on site with the Sofia SARS Antigen FIA test. The results of the two tests will then be compared.
  These samples will not be collected for further research.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
assessment Vs gold standard | Up to 35 positive PCR
  PCR results and Ct values for specimens tested are collected and compared with Sofia results.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre de dépistage - CHRU BREST, Brest
  - CHRU de brest, Brest

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three month and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.